CLINICAL TRIAL: NCT06447311
Title: Assessing the Clinical Efficacy of Hyaluronic Acid Hydrogel in Papilla Augmentation: A Clinical Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr R Viswa Chandra (Other)
Responsible Party: Sponsor-Investigator, Dr R Viswa Chandra, PROFFESSOR AND HEAD OF THE DEPARTMENT, SVS Institute of Dental Sciences
Organization: SVS Institute of Dental Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVSInstituteDS4
Record Dates: First submitted 2024-05-20; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Gingival Destruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): In Test group, the prepared Hyaluronic acid gel will be injected using a syringe into the defect site.
  Interventions: Other: Hyaluronic acid gel
- Control group (Placebo Comparator): In Control group, saline placebo gel will be injected into the defect site using a syringe.
  Interventions: Other: Hyaluronic acid gel

INTERVENTIONS:
Other: Hyaluronic acid gel — Hyaluronic acid is involved in tissue repair and wound healing by stimulating cell proliferation, migration and interaction with several growth factors. Furthermore, HA has a crucial role in space-filling owing to its hygroscopic nature.

SUMMARY:
The aim of this study is to evaluate the effect of hyaluronic acid gel in papilla augmentation.

DETAILED DESCRIPTION:
Assessing the clinical efficacy of Hyaluronic acid hydrogel in papilla augmentation: A clinical study.

In Test group, Hyaluronic acid hydrogel will be injected using a syringe into the interdental papillary deficiency site.

In Control group, saline placebo gel will be injected into the interdental papillary deficiency site using a syringe.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking patients aged above 18 years.
2. Have at least one site with interdental papilla recession in the anterior region (central incisors, lateral incisors and canines) of the maxillary or mandibular jaws.
3. Class I or Class II papillary recession.
4. The distance from the contact point to alveolar bone crest ≥5mm.
5. No active periodontal diseases and good oral hygiene.

Exclusion Criteria:

1. spacing or crowding between the teeth to be treated,
2. abnormal tooth shape,
3. systemic diseases such as diabetes mellitus, hypertension or
4. conditions that alter the outcome of periodontal therapy.
5. Pregnant and lactating women and
6. tobacco users

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of papilla augmentation | Baseline to 6 months
  Assessment of the empty space left by the receding interdental papilla will be measured using UNC-15 probe at baseline and post-operatively at 3 and 6 months.

SECONDARY OUTCOMES:
Assessment of plaque | baseline ,3months,6months
  Assessment of plaque (PI) - according to Turesky modification of Quigley and Hein Plaque Index, 1970
Assessment of gingiva | baseline ,3months,6months
  Gingival index (GI) - according to Loe H and Silness P, 1963

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute of dental sciences, Mahbūbnagar, Telangana, India

IPD SHARING:
Plan to Share IPD: No